CLINICAL TRIAL: NCT04833855
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose-Ranging, Phase 2b Study to Evaluate Efficacy and Safety of Tezepelumab for the Treatment of Chronic Spontaneous Urticaria
Brief Title: Study to Evaluate Tezepelumab in Adults With Chronic Spontaneous Urticaria
Acronym: INCEPTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20190194
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CSU
MeSH Terms: conditions — Chronic Urticaria | interventions — tezepelumab; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1: Omalizumab (Active Comparator): Participants naive to anti-IgE therapies will receive omalizumab.
  Interventions: Biological: Omalizumab
- Group 2: Placebo (Placebo Comparator): Participants naive to anti-IgE therapies will receive a placebo.
  Interventions: Biological: Placebo
- Group 3: Tezepelumab Dose 1 (Experimental): Participants naive to anti-IgE therapies will receive tezepelumab.
  Interventions: Biological: Tezepelumab Dose 1
- Group 4: Tezepelumab Dose 2 (Experimental): Participants naive to anti-IgE therapies will receive tezepelumab.
  Interventions: Biological: Tezepelumab Dose 2
- Group 5: Placebo (Placebo Comparator): Participants previously treated with anti-IgE therapies will receive a placebo.
  Interventions: Biological: Placebo
- Group 6: Tezepelumab Dose 1 (Experimental): Participants previously treated with anti-IgE therapies will receive tezepelumab.
  Interventions: Biological: Tezepelumab Dose 1
- Group 7: Tezepelumab Dose 2 (Experimental): Participants previously treated with anti-IgE therapies will receive tezepelumab.
  Interventions: Biological: Tezepelumab Dose 2

INTERVENTIONS:
Biological: Tezepelumab Dose 1 — Subcutaneous injection.
  Other Names: AMG 157
  Arms: Group 3: Tezepelumab Dose 1; Group 6: Tezepelumab Dose 1
Biological: Tezepelumab Dose 2 — Subcutaneous injection.
  Other Names: AMG 157
  Arms: Group 4: Tezepelumab Dose 2; Group 7: Tezepelumab Dose 2
Biological: Omalizumab — Subcutaneous injection.
  Other Names: Xolair
  Arms: Group 1: Omalizumab
Biological: Placebo — Subcutaneous injection.
  Arms: Group 2: Placebo; Group 5: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of tezepelumab on improvement in the Urticaria Activity Score over 7 days (UAS7).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male and female participants ≥ 18 years and ≤ 80 years of age at the time of screening.
* Chronic spontaneous urticaria (CSU) diagnosis for ≥ 6 months at the time of screening.
* CSU inadequately controlled by second generation H1-antihistamines (sgAH) at enrollment, as defined by all of the following:
* The presence of itch and hives for >= 6 consecutive weeks at any time prior to screening visit 2
* Failure to respond to an sgAH (up to 4 times the approved dose)
* Urticaria Activity Score over 7 days (UAS7) (range 0-42) >= 16 and Hives Severity Score over 7 days (HSS7) (range 0-21) >= 8 during the 7 days prior to enrollment
* Participant with CSU who discontinued, is intolerant to, or was an inadequate responder to anti-IgE therapies despite being treated with omalizumab 300 mg every 4 weeks (Q4W) for 6 months or higher doses of omalizumab > 2 months or another anti-IgE therapy. Note: This criterion is only applicable for anti-IgE-experienced participants.
* Participant willing and able to complete a daily symptom eDiary for the duration of the study and adhere to the study visit schedules.
* Subject must have been on a sgAH at approved or increased doses (up to 4x the approved dose) for treatment of CSU for at least 3 consecutive days immediately prior to the day -14 screening visit (screening visit 2) and must have documented current use on the day of screening visit 1

Exclusion Criteria:

Disease related, including but not limited to:

* Urticaria is solely due to inducible urticaria
* Active dermatologic diseases (or conditions) other than chronic urticaria, with urticaria wheals or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to C1 inhibitor deficiency)
* Any other active skin disease associated with chronic itching that might influence, in the investigator's opinion, the study evaluations and results (eg, atopic dermatitis, dermatitis herpetiformis, senile pruritus, etc.)
* History of a clinically significant infection within 28 days prior to day 1 that, in the opinion of the investigator or medical monitor, might compromise the safety of the participant in the study, interfere with evaluation of the investigational product, or reduce the participants ability to participate in the study.
* Evidence of active tuberculosis (TB) (in the opinion of the investigator), either treated or untreated, or a positive purified protein derivative (PPD) or QuantiFERON-TB Gold Plus (QFT-Plus) test for TB during screening.
* History of malignancy, except for basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy ≥ 12 months prior to screening or other malignancies treated with apparent success with curative therapy ≥ 5 years prior to screening visit 1.
* Subject is unable to complete an electronic patient diary or complete questionnaires, or does not meet the required level of compliance with the eDiary during the 14 days sgAH stabilization period

Other medical conditions

* History or evidence of severe depression, schizophrenia, previous suicide attempts, or suicidal ideation.

Prior/concomitant therapy, including but not limited to:

* Treatment with any biologic products (eg, omalizumab, ligelizumab) within 4 months or 5 half-lives (whichever is longer) prior to screening visit 1
* Routine (daily or every other day for 5 or more consecutive days) use of systemic corticosteroids, systemic hydroxychloroquine, methotrexate, cyclosporine A, cyclophosphamide, tacrolimus, azathioprine, and mycophenolate mofetil within 30 days prior to screening visit 1.
* Major surgery within 8 weeks prior to screening visit 1 or planned inpatient surgery or hospitalization during the study period.
* Receipt of Ig or blood products within 30 days prior to screening visit 1.
* Vaccination with a live or attenuated vaccine within 30 days prior to screening visit 1. Receipt of COVID-19 vaccines and inactive/killed vaccinations (eg, inactive influenza) are allowed, provided the vaccinations are not administered within 7 days before or after any study dosing visit.
* Known hypersensitivity, including severe hypersensitivity reactions and/or history of anaphylactic shock, to any of the products or components to be administered during dosing or to products of similar chemical classes (ie, to murine, chimeric, or human antibodies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (81):
- United States (25):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - First OC Dermatology, Fountain Valley, California
  - Avance Clinical Trials, Laguna Niguel, California
  - Jonathan Corren MD Inc, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Asthma and Allergy Associates PC, Colorado Springs, Colorado
  - The Community Research of South Florida, Miami Lakes, Florida
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - Bluegrass Allergy Care, Lexington, Kentucky
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - David Fivenson MD Professional Liability Company, Ann Arbor, Michigan
  - Clarkston Skin Research, Clarkston, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Bernstein Clinical Research Center LLC, Cincinnati, Ohio
  - Aventiv Research Inc, Dublin, Ohio
  - Clinical Partners LLC, Johnston, Rhode Island
  - The Allergy Asthma and Sinus Center, East Tennessee Center for Clinical Research, Knoxville, Tennessee
  - Suzanne Bruce and Associates, Houston, Texas
  - Cutis Wellness Dermatology and Dermatopathology, PLLC, Laredo, Texas
- Canada (9):
  - Dermatology Research Institute Incorporated, Calgary, Alberta
  - Brunswick Dermatology Centre, Fredericton, New Brunswick
  - LEADER Research, Hamilton, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - Cheema Research Incorporated, Mississauga, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario
  - Allergy Research Canada Incorporated, Niagara Falls, Ontario
  - Gordon Sussman Clinical Research Incorporated, North York, Ontario
  - Clinique Spécialisée en Allergie de la Capitale, Québec, Quebec
- France (5):
  - Centre Hospitalier Universitaire de Brest - Hôpital Morvan, Brest
  - Centre Hospitalier Universitaire de Grenoble - Hopital Nord Michallon, Grenoble
  - Hôpital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire Archet 2, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (3):
  - *Charité*, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - Johannes Gutenberg Universitaet Mainz, Mainz
- Greece (5):
  - Laiko General Hospital of Athens, Athens
  - Sotiria General Hospital, Athens
  - Attikon University General Hospital of Athens, Athens
  - Andreas Syggros Hospital, Athens
  - George Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Italy (6):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Fondazione Policlinico Tor Vergata, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Japan (9):
  - Fujita Health University Bantane Hospital, Nagoya, Aichi-ken
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Takagi Dermatological Clinic, Obihiro-shi, Hokkaido
  - Kosugi Dermatology Clinic, Kawasaki-shi, Kanagawa
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Osaka Habikino Medical Center, Habikino-shi, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai-shi, Osaka
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
- Poland (8):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - AMICARE z ograniczona odpowiedzialnoscia spolka komandytowa, Lodz
  - SPZOZ Centralny Szpital Kliniczny, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - Kliniczny Szpital Wojewodzki nr 1 im Fryderyka Chopina, Rzeszów
  - Klinika Osipowicz and Turkowski Spzoo Opieka Wielospecjalistyczna Osipowicz and Turkowski, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- South Korea (6):
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ajou University Hospital, Suwon-si, Gyeonggi-do
- Spain (5):
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] McLaren J, Chon Y, Gorski KS, Bernstein JA, Corren J, Hayama K, Jain V, Lima H, Sofen H, Ponnarambil S, Molfino NA, Maurer M. Tezepelumab for the treatment of chronic spontaneous urticaria: Results of the phase 2b INCEPTION study. J Allergy Clin Immunol. 2025 Jun;155(6):1945-1956. doi: 10.1016/j.jaci.2025.01.045. Epub 2025 Feb 14. PMID 39956278
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 56 study centers in Japan, Republic of Korea, France, Germany, Greece, Italy, Poland, Spain, Canada, and the United States, and participated from 15 April 2021 to 13 April 2023.
Pre-assignment Details: Participants with chronic spontaneous urticaria (CSU) and symptomatic despite treatment with second generation H1-antihistamines (sgAH) were randomized based on if they were previously treated with anti-immunoglobulin E (IgE) therapies or were anti-IgE naïve.
Groups:
- Placebo: Participants with and without previous anti-IgE therapy experience were randomized to receive placebo subcutaneously (SC) every 2 weeks (Q2W) for 16 weeks.
  Participants maintained a stable dose of sgAH as background medication from screening Visit 2 (Day -14) to the end of the Safety Follow-up Period (up to Week 32).
- Omalizumab 300 mg SC Q4W: Participants without previous anti-IgE experience were randomized to receive omalizumab 300 mg SC every 4 weeks (Q4W) for 16 weeks. Participants received placebo SC at intervening study visits to ensure all participants received an injection Q2W.
  Participants maintained a stable dose of sgAH as background medication from screening Visit 2 (Day -14) to the end of the Safety Follow-up Period (up to Week 32).
- Tezepelumab 210 mg SC Q4W: Participants with and without previous anti-IgE therapy experience were randomized to receive tezepelumab 210 mg SC Q4W for 16 weeks. Participants received placebo SC at intervening study visits to ensure all participants received an injection Q2W.
  Participants maintained a stable dose of sgAH as background medication from screening Visit 2 (Day -14) to the end of the Safety Follow-up Period (up to Week 32).
- Tezepelumab 420 mg SC Q2W: Participants with and without previous anti-IgE therapy experience were randomized to receive tezepelumab 420 mg SC Q2W for 16 weeks.
  Participants maintained a stable dose of sgAH as background medication from screening Visit 2 (Day -14) to the end of the Safety Follow-up Period (up to Week 32).
Period: Overall Study
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Started | 48 | 31 | 52 | 52
Completed | 43 | 29 | 45 | 48
Not Completed | 5 | 2 | 7 | 4
Not completed — Decision by sponsor | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 2
Not completed — Protocol specified criteria | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants with and without previous anti-IgE therapy experience were randomized to receive placebo SC Q2W for 16 weeks.
  Participants maintained a stable dose of sgAH as background medication from screening Visit 2 (Day -14) to the end of the Safety Follow-up Period (up to Week 32).
- Omalizumab 300 mg SC Q4W: Participants without previous anti-IgE experience were randomized to receive omalizumab 300 mg SC Q4W for 16 weeks. Participants received placebo SC at intervening study visits to ensure all participants received an injection Q2W.
  Participants maintained a stable dose of sgAH as background medication from screening Visit 2 (Day -14) to the end of the Safety Follow-up Period (up to Week 32).
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W | Total
Number analyzed (Participants) | 48 | 31 | 52 | 52 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (15.2) | 39.8 (13.1) | 45.0 (14.7) | 42.9 (14.5) | 42.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 23 | 35 | 39 | 134
  Male | 11 | 8 | 17 | 13 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 6 | 14
  Not Hispanic or Latino | 45 | 29 | 49 | 46 | 169
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18 | 12 | 16 | 14 | 60
  Black or African American | 1 | 2 | 2 | 2 | 7
  Multiple | 0 | 0 | 0 | 1 | 1
  White | 29 | 17 | 34 | 34 | 114
  Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urticaria Activity Score Over 7 Days (UAS7) at Week 16
Description: The UAS is a CSU-specific patient-reported outcome measure with 2 components: Hives Severity Score (HSS) for number of wheals and an Itch Severity Score (ISS) for itch intensity, and are each scored from 0 (no wheals, no itch) to 3 (>50 wheals, severe itch) for the previous 24 hours. The HSS and ISS are combined to give a daily UAS ranging from 0 to 6. The sum of the daily UAS over a 7-day period provides the UAS7, from 0 (no symptoms) to 42 (severe urticaria). The least squares mean (LSM) estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline UAS7, treatment, study week and the interaction between treatment and study week. A negative change from baseline indicates an improvement in urticaria activity.
Time Frame: Baseline and Week 16
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
score on a scale | -13.6 (1.6) | -18.4 (2.0) | -13.5 (1.6) | -14.7 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 210 mg SC Q4W; Test type: Superiority; p = 0.99, Repeated measure model — Nominal p-value; Model parameters: stratification factor (prior anti-IgE status), baseline UAS7, treatment, study week, interaction between treatment and study week; LSM difference = 0.0, 95% CI 2-sided [-4.3 to 4.4], Standard Error of Mean 2.2 — Tezepelumab 210 mg SC Q4W - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 420 mg SC Q2W; Test type: Superiority; p = 0.60, Repeated measure model — Nominal p-value; [statistical method as in outcome 1, analysis 1]; LSM difference = -1.1, 95% CI 2-sided [-5.4 to 3.1], Standard Error of Mean 2.2 — Tezepelumab 420 mg SC Q2W - Placebo

2. Secondary Outcome: Change From Baseline in ISS Over 7 Days (ISS7) at Week 16
Description: The ISS is a component of the UAS, a CSU-specific patient-reported outcome measure and assessed itch intensity, with daily scores ranging from 0 (no itch) to 3 (severe itch) for the previous 24 hours. The sum of daily ISS over a 7-day period provides the ISS7, from 0 (no symptoms) to 21 (severe itch). The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline ISS7, treatment, study week and the interaction between treatment and study week. A negative change from baseline indicates an improvement in urticaria activity.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
score on a scale | -7.7 (0.8) | -9.6 (1.0) | -7.3 (0.8) | -8.0 (0.8)

3. Secondary Outcome: Change From Baseline in HSS Over 7 Days (HSS7) at Week 16
Description: The HSS is a component of the UAS, a CSU-specific patient-reported outcome measure and assessed the number of wheals, with daily scores ranging from 0 (no wheals) to 3 (>50 wheals) for the previous 24 hours. The sum of daily HSS over a 7-day period provides the HSS7, from 0 (no symptoms) to 21 (severe wheals). The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline HSS7, treatment, study week and the interaction between treatment and study week. A negative change from baseline indicates an improvement in urticaria activity.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
score on a scale | -5.8 (0.8) | -8.8 (1.1) | -6.3 (0.8) | -6.7 (0.8)

4. Secondary Outcome: Number of Participants With a UAS7 of ≤ 6 (Minimal Residual Disease) at Week 16
Description: The sum of the daily UAS over a 7-day period provides the UAS7, from 0 (no symptoms) to 42 (severe urticaria). Minimal residual disease in UAS7 was defined as a score ≤ 6 and indicates well-controlled urticaria and a good response to treatment.
Time Frame: Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product. Participants with observed data are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 39 | 25 | 39 | 48
Participants | 8 | 14 | 10 | 13

5. Secondary Outcome: Number of Participants With a Change From Baseline in UAS7 of ≤ -10 (Minimal Important Difference)
Description: The sum of the daily UAS over a 7-day period provides the UAS7, from 0 (no symptoms) to 42 (severe urticaria). Minimal important difference in UAS7 was defined as a change from baseline of ≤ -10.
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 39 | 25 | 39 | 48
Participants | 28 | 20 | 27 | 32

6. Secondary Outcome: Number of Participants With a UAS7 = 0 at Week 16 (Complete Response)
Description: The sum of the daily UAS over a 7-day period provides the UAS7, from 0 (no symptoms) to 42 (severe urticaria). A complete response was defined as UAS7 = 0 at Week 16.
Time Frame: Week 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 39 | 25 | 39 | 48
Participants | 4 | 11 | 7 | 5

7. Secondary Outcome: Number of Participants With ISS7 = 0 at Week 16 (Complete Resolution)
Description: The sum of daily ISS over a 7-day period provides the ISS7, from 0 (no symptoms) to 21 (severe itch). An ISS7 = 0 indicates a complete resolution of itch.
Time Frame: Week 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 39 | 25 | 39 | 48
Participants | 4 | 12 | 7 | 9

8. Secondary Outcome: Number of Participants With a Change From Baseline in ISS7 of ≤ -5 (Minimal Important Difference)
Description: The sum of daily ISS over a 7-day period provides the ISS7, from 0 (no symptoms) to 21 (severe itch). Minimal important difference in ISS7 was defined as a change from baseline of ≤ -5.
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 39 | 25 | 39 | 48
Participants | 29 | 20 | 28 | 34

9. Secondary Outcome: Number of Participants With HSS7 = 0 at Week 16 (Complete Resolution)
Description: The sum of daily HSS over a 7-day period provides the HSS7, from 0 (no symptoms) to 21 (severe wheals). An HSS7 = 0 indicates a complete resolution of hives.
Time Frame: Week 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 39 | 25 | 39 | 48
Participants | 6 | 11 | 8 | 6

10. Secondary Outcome: Number of Participants With a Change From Baseline in HSS7 of ≤ -5.5 (Minimal Important Difference)
Description: The sum of daily HSS over a 7-day period provides the HSS7, from 0 (no symptoms) to 21 (severe wheals). Minimal important difference in HSS7 was defined as a change from baseline of ≤ -5.5.
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 39 | 25 | 39 | 48
Participants | 23 | 19 | 24 | 31

11. Secondary Outcome: Change From Baseline in Weekly Sleep Interference Score (SIS7) at Week 16
Description: The SIS is part of the Urticaria Patient Daily Diary and was assessed by the participant using the electronic diary once daily in the morning. Participants scored sleep interference on a scale of 0 (no interference) to 3 (substantial, woke up often, severe interference with sleep). The SIS7 was a sum of the daily scores over 7 days ranging from 0 to 21. The LSM estimates were based on the repeated measure model with stratification factor (prior anti-IgE status), baseline SIS7, treatment, study week and the interaction between treatment and study week. A negative change from baseline indicates an improvement in sleep interference.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
score on a scale | -8.4 (0.7) | -6.5 (0.9) | -7.4 (0.7) | -7.8 (0.7)

12. Secondary Outcome: Change From Baseline in Weekly Sleep Quality Score (SQS7): Sum of Daily SQS at Week 16
Description: The SQS was assessed by the participant through 3 questions relating to falling asleep (Q1), wakefulness (Q2), and feeling rested in the morning (Q3). The sum of the 3 daily sleep quality items over 7 days, ranged from 0 (good quality sleep) to 63 (poor quality sleep). The LSM estimates were based on the repeated measure model with stratification factor (prior anti-IgE status), baseline SQS7 - sum of SQS, treatment, study week and the interaction between treatment and study week. A negative change from baseline indicates an improvement in sleep quality.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
score on a scale | -19.5 (1.8) | -16.7 (2.3) | -18.3 (1.7) | -17.1 (1.6)

13. Secondary Outcome: Change From Baseline in SQS7: Sum of Average Daily Q1 - Q3 at Week 16
Description: The SQS was assessed by the participant through 3 questions relating to falling asleep (Q1), wakefulness (Q2), and feeling rested in the morning (Q3). The sum of average daily Q1 - Q3 score was generated by averaging 3 daily sleep quality items and then summing the daily average over 7 days with a score ranging from 0 (good quality sleep) to 21 (poor quality sleep) (sum of the average daily Q1 - Q3). The LSM estimates were based on the repeated measure model with stratification factor (prior anti-IgE status), baseline SQS7 - sum of average daily Q1 - Q3, treatment, study week and the interaction between treatment and study week. A negative change from baseline indicates an improvement in sleep quality.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
score on a scale | -6.5 (0.6) | -5.6 (0.8) | -6.1 (0.6) | -5.7 (0.5)

14. Secondary Outcome: Change From Baseline in Urticaria Control Test (UCT) Score at Week 16
Description: The UCT assesses disease control in participants with CSU through a retrospective validated scoring system, evaluating the physical symptoms of chronic urticaria (itch, hives and/or angioedema) and the effectiveness of treatment over 4 weeks. It consists of 4 questions with 5 answer options, scored from 0 to 4, and the UCT score is the sum of all 4 questions, with total score ranging from 0 (no control) to 16 (complete control). A score of ≥ 12 indicates well-controlled urticaria and a score of ≤ 11 points indicates poor disease control. A positive change from baseline indicates an improvement in disease control. The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline UCT score, treatment, study week and the interaction between treatment and study week.
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 46 | 29 | 48 | 49
score on a scale | 4.1 (0.6) | 6.3 (0.8) | 4.9 (0.6) | 5.9 (0.6)

15. Secondary Outcome: Change From Baseline in Weekly Angioedema Activity Score (AAS7) at Week 16
Description: The AAS is a 5-item patient-reported outcome measure used to determine angioedema activity. Participants retrospectively documented the presence or absence of angioedema in the past 24 hours, and the AAS daily score ranged from 0 to 15 points, assessing 5 key factors when angioedema is present, including duration, physical discomfort, impact on daily activities, impact on appearance, and overall severity). The daily AAS scores are summed for 7 days to form the AAS7 with a range of 0 (not present) to 105 (most severe angioedema activity). Negative changes from baseline indicate an improvement in angioedema activity. The LSM estimates were based on the repeated measure model with stratification factor (prior anti-IgE status), baseline AAS7, treatment, study week and the interaction between treatment and study week.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
score on a scale | -19.0 (2.7) | -18.7 (3.5) | -20.8 (2.7) | -15.6 (2.5)

16. Secondary Outcome: Number of Cumulative Weeks That Participants Achieved AAS7 = 0 at Week 16 (Angioedema Occurrence Free)
Description: The AAS is a 5-item patient-reported outcome measure used to determine angioedema activity. Participants retrospectively documented the presence or absence of angioedema in the past 24 hours, and the AAS daily score ranged from 0 to 15 points, assessing 5 key factors when angioedema is present, including duration, physical discomfort, impact on daily activities, impact on appearance, and overall severity). The daily AAS scores are summed for 7 days to form the AAS7 with a range of 0 (not present) to 105 (most severe angioedema activity). Angioedema occurrence free was defined as AAS7 = 0.
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 40 | 26 | 44 | 37
weeks | 10.8 (5.2) | 11.3 (4.9) | 9.9 (5.8) | 11.5 (5.4)

17. Secondary Outcome: Change From Baseline in the Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) at Week 16
Description: The CU-Q2oL is a 23-item, self-reported urticaria-specific measure to evaluate 6 dimensions of quality of life (QoL): pruritus, impact on life activities, sleep problems, limitations, looks, and swelling. The total score is transformed to a linear scale of 0 to 100 with a higher CU-Q2oL score indicating a higher QoL impairment. A negative change from baseline indicates an improvement in QoL. The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline CU-Q2oL score, treatment, study week and the interaction between treatment and study week.
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 44 | 25 | 41 | 44
score on a scale | -19.6 (2.1) | -19.8 (2.8) | -19.3 (2.2) | -18.7 (2.1)

18. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item, participant-completed, health-related QoL assessment with content specific to those with dermatology conditions. The DLQI evaluates participant perceptions including dermatology-related symptoms and feelings, impacts on daily activities, leisure, work or school, personal relationships, and side effects of treatment. The recall period was 1 week. The DLQI total score ranges from 0 to 30 with a higher score indicating a greater QoL impairment. A negative change from baseline indicates an improvement in QoL. The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline DLQI score, treatment, study week and the interaction between treatment and study week.
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 44 | 25 | 41 | 44
score on a scale | -7.4 (0.9) | -7.3 (1.2) | -7.0 (0.9) | -7.0 (0.9)

19. Secondary Outcome: Change From Baseline in the Angioedema Quality of Life Questionnaire (AE-QoL) at Week 16
Description: The AE-QoL is a validated angioedema QoL questionnaire for participants with angioedema. It consists of 17 questions evaluating 4 domains including functioning, fatigue/mood, fear/shame, and food with a recall period of 4 weeks. The total score is transformed to a linear scale ranging from 0 to 100, with a higher score indicating a worse impairment in QoL. A negative change from baseline indicates an improvement in QoL. The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline AE-QoL score, treatment, study week and the interaction between treatment and study week.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product. Participants with angioedema presence at baseline and at least 1 non-missing AE-QoL record were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 20 | 7 | 15 | 16
score on a scale | -29.2 (6.0) | -24.1 (10.9) | -24.6 (6.4) | -13.1 (7.4)

20. Secondary Outcome: Change From Baseline in the Angioedema Control Test (AECT) Score at Week 16
Description: The AECT is a patient-reported outcome measure to evaluate disease control in the domains of signs and symptoms, QoL, anxiety/fear, and effectiveness of therapy. The total AECT score ranges from 0 to 16, with higher scores indicating well-controlled disease. A positive change from baseline indicates an improvement in angioedema control. The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline AECT score, treatment, study week and the interaction between treatment and study week.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product. Participants with angioedema presence at baseline and at least 1 non-missing AECT record were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 20 | 7 | 15 | 16
score on a scale | 4.2 (1.2) | 3.9 (2.2) | 4.6 (1.3) | 2.3 (1.5)

21. Secondary Outcome: Number of Participants With an AECT Score = 16 at Week 16 (Complete Control)
Description: The total AECT score ranges from 0 to 16, with higher scores indicating better controlled disease. Complete control was defined as AECT score = 16.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product. Participants with observed data at Week 16 and angioedema presence at baseline and at least 1 non-missing AECT record were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 15 | 5 | 14 | 14
Participants | 3 | 2 | 0 | 1

22. Secondary Outcome: Change From Baseline in the Work Productivity and Activity Impairment Questionnaire: Chronic Urticaria (WPAI-CU) Score at Week 16
Description: The WPAI-CU is a questionnaire that assesses the impact of an intervention on work productivity, evaluating 4 areas including absenteeism, presenteeism, work productivity loss, and activity impairment over the past 7 days. Each of the areas is scored separately as a percentage, ranging from 0 to 100, with higher numbers indicating greater impairment and less productivity. A negative change from baseline indicates an improvement. The LSM estimates are based on the repeated measure model with stratification factor (prior anti-IgE status), baseline WPAI-CU score, treatment, study week and the interaction between treatment and study week.
Time Frame: Baseline and Week 16
Population: The FAS included all randomized participants who received at least 1 dose of investigational product. Participants with observed data were included for each question.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 44 | 25 | 41 | 44
score on a scale
  Absenteeism: number analyzed (Participants) | 33 | 20 | 28 | 26
  Absenteeism | -4.7 (2.5) | 0.3 (3.0) | -7.5 (2.5) | -2.3 (2.7)
  Presenteeism: number analyzed (Participants) | 32 | 19 | 27 | 24
  Presenteeism | -19.9 (5.2) | -18.3 (6.6) | -20.3 (5.3) | -17.8 (5.7)
  Work productivity loss: number analyzed (Participants) | 32 | 19 | 27 | 24
  Work productivity loss | -20.0 (5.4) | -13.3 (6.7) | -23.5 (5.5) | -17.5 (5.9)
  Activity impairment | -28.5 (4.2) | -30.3 (5.6) | -27.2 (4.3) | -24.1 (4.1)

23. Secondary Outcome: Number of Cumulative Days of sgAH Rescue Medication Use From Baseline to Week 16
Description: Participants recorded any need of sgAH rescue medication in their daily electronic diary.
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 22 | 19 | 31 | 25
days | 49.5 (39.0) | 31.6 (42.7) | 46.1 (39.3) | 32.7 (33.4)

24. Secondary Outcome: Serum Concentration of Tezepelumab
Description: The lower limit of quantification was 10 ng/mL, and values below this limit were set to zero.
Time Frame: Week 1 pre-dose, Weeks 2, 4, 8, 12, 16, 24, and 32
Population: The pharmacokinetic analysis set included participants who received tezepelumab and had at least 1 sample with a measurable serum concentration. Participants with data available at each time point are included.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 51 | 52
µg/mL
  Week 1 | 0.00 (0.00) | 0.00 (0.00)
  Week 2: number analyzed (Participants) | 51 | 48
  Week 2 | 20.1 (6.93) | 41.3 (12.4)
  Week 4: number analyzed (Participants) | 46 | 47
  Week 4 | 14.2 (5.78) | 71.3 (20.8)
  Week 8: number analyzed (Participants) | 41 | 43
  Week 8 | 21.2 (8.54) | 101 (30.5)
  Week 12: number analyzed (Participants) | 38 | 43
  Week 12 | 24.8 (9.67) | 123 (44.1)
  Week 16: number analyzed (Participants) | 39 | 41
  Week 16 | 27.1 (10.7) | 136 (43.4)
  Week 24: number analyzed (Participants) | 37 | 39
  Week 24 | 6.95 (5.65) | 37.3 (21.1)
  Week 32: number analyzed (Participants) | 40 | 42
  Week 32 | 1.73 (1.73) | 11.0 (10.8)

25. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with study treatment. TEAEs were AEs that started on or after the first dose of investigational product up to the end of study (Week 32). A serious AE (SAE) was defined as any untoward medical occurrence that met at least 1 of the following serious criteria: immediately life-threatening, required hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or other medically important serious event.
Time Frame: Day 1 Week 1 to Week 32, up to 32 weeks
Population: The safety analysis set consisted of all randomized participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
Number analyzed (Participants) | 48 | 31 | 52 | 52
Participants
  TEAEs | 23 | 24 | 29 | 28
  SAEs | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrolment to the end of study visit, up to 38 weeks. SAEs and other AEs were collected from Day 1 up to Week 32, up to 32 weeks.
Arm/Group | Placebo | Omalizumab 300 mg SC Q4W | Tezepelumab 210 mg SC Q4W | Tezepelumab 420 mg SC Q2W
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/31 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/31 | 1/52 | 0/52
Other Adverse Events (participants affected / at risk) | 14/48 | 7/31 | 19/52 | 20/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Omalizumab 300 mg SC Q4W (N=31) | Tezepelumab 210 mg SC Q4W (N=52) | Tezepelumab 420 mg SC Q2W (N=52)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Omalizumab 300 mg SC Q4W (N=31) | Tezepelumab 210 mg SC Q4W (N=52) | Tezepelumab 420 mg SC Q2W (N=52)
Injection site pain (General disorders) | 1 | 0 | 4 | 1
Pyrexia (General disorders) | 1 | 3 | 3 | 2
COVID-19 (Infections and infestations) | 3 | 2 | 8 | 5
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Headache (Nervous system disorders) | 2 | 1 | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT04833855/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT04833855/SAP_001.pdf